CLINICAL TRIAL: NCT07059182
Title: Phase 1 Trial to Assess Safety and Tolerability of a Single Dose of Streptococcus Pneumoniae Whole-Cell (wSp) Vaccine in Healthy Adults
Brief Title: Safety Study of a Single Dose of Pneumococcal Whole-Cell Vaccine in Healthy Adults
Acronym: STREPTO VAC I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: wSp-US-1.05AOM
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: PREVENTION OF INVASIVE PNEUMOCOCCAL DISEASE; Prevention of Pneumococcal-induced Acute Otitis Media
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1x 1 mg wSp vaccine (Experimental): The study product, wSp vaccine, will be supplied as single-dose glass vials in normal saline (0.9% sodium chloride) at 1 mg protein/0.5 mL, with aluminium hydroxide at 1.2 mg elemental Al/mL. 0.5 mL of study product will be administered in the participant's deltoid as an intramuscular injection.
  Interventions: Biological: Inactivated whole-cell Streptococcus pneumoniae vaccine
- Placebo (Placebo Comparator): Placebo will consist of normal saline (0.9% sodium chloride). 0.5 mL of placebo will be administered in the participant's deltoid as an intramuscular injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Inactivated whole-cell Streptococcus pneumoniae vaccine — Single intramuscular injection of 1 mg protein/0.5 mL wSp vaccine
  Other Names: Streptococcus pneumoniae Whole Cell Vaccine (SPWCV); wSp vaccine
  Arms: 1x 1 mg wSp vaccine
Drug: Placebo — Single intramuscular injection of 0.5 mL placebo
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if whole-cell Streptococcus pneumoniae (wSp) vaccination is safe and tolerated in healthy adults. The main aim is to evaluate the safety and tolerability of wSp vaccine.

Researchers will compare wSp vaccinated participants with placebo-treated participants.

Participants will be administered once with 1mg wSp vaccine or placebo. After dosing, they will be followed up for 30 days. In addition to the screening and enrollment visits, each participant will come to the study site for scheduled study visits on Days 14 and 30 to undergo study evaluations and measurements and to monitor safety. Each participant also will receive scheduled phone calls on Days 3 and 7 to monitor safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged > 18 and < 49 years at screening.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2, with a maximum body weight of 120 kg at screening.
* Good general health, without significant medical illness or abnormal physical examination, or laboratory findings per PI discretion.
* If female, not breastfeeding, not pregnant, and not planning pregnancy during study period.
* If female of child-bearing potential, willing to use acceptable method of contraception.
* Willing and able to comply with all study activities, assessments, and restrictions through 30 days of follow-up. Willing and able to be contacted reliably by phone, and willing for the study team to record phone voice messages as needed.
* Provided written informed consent to participate in the clinical trial before any study-related activities are carried out and, in the PI's opinion, must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.

Exclusion Criteria:

In addition to meeting the inclusion criteria, individuals will be excluded from this trial if they meet any of the following exclusion criteria:

* History or presence of clinically significant medical condition or disease, including (but not limited to) clinically significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, hematologic, immunologic, oncologic, rheumatologic, dermatologic, neurological or psychiatric disease.
* History of known invasive pneumococcal disease.
* History of congenital or acquired immunodeficiency.
* Any acute illness within 72 hours prior to randomization.
* Abnormal vital sign(s) or laboratory test result(s) deemed clinically relevant, as determined by the PI.
* Known allergy or previous anaphylaxis to any components of the study product or contraindication to intramuscular (IM) injection (e.g., history of bleeding disorder).
* Previous enrollment in this trial or received other investigational vaccines, drugs, or products within the past 12 weeks, or intend to participate in another clinical trial during the duration of this trial.
* Received any vaccine within the past 4 weeks.
* Received any immunomodulating or immunosuppressive agent or medicine, including over-the-counter, herbal and prescription drugs and supplements within the past 12 weeks or anticipate needing within the study period.
* Received blood or blood products within the past 12 weeks or anticipate needing within the study period.
* Current use of over the counter or prescription drugs of known hepatotoxicity.
* Current or history of alcohol or drug dependence or abuse.
* Any condition (medical, psychiatric, or behavioral) that in the opinion of the PI, would increase the participant's health risks in study participation or would increase the risk of not achieving the study's objectives.
* Unable or unwilling to provide adequate informed consent.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability outcome | within 7 days post-vaccination//through Day 30
  Occurrence and severity of local reactogenicity (injection site pain, tenderness, redness, swelling, itching, local lymphadenopathy) and systemic reactogenicity (headache, muscle pain, fever, nausea, vomiting, excessive fatigue, and diarrhea) within 7 days post-vaccination.
  Occurrence, severity, and relatedness of solicited AEs and SAEs through Day 30.
  Occurrence, severity, and relatedness of unsolicited AEs and SAEs through Day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Clinical Research, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT07059182/ICF_000.pdf